CLINICAL TRIAL: NCT01291940
Title: The Effects of Emollient Therapy on the Skin Barrier Function
Brief Title: The Effects of Emollient Therapy on the Skin Barrier
Acronym: EES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Eric Simpson, MD, MCR, Oregon Health and Science University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Emollient Evaluation Study
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Petrolatum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pediatric Moisturizer Intervention (Experimental): Apply one of four moisturizers to one arm daily for four weeks.
  Interventions: Other: Pediatric Moisturizer
- Adult Moisturizer Intervention (Experimental): Apply moisturizer to one arm once a day for four weeks.
  Interventions: Other: Adult Moisturizer
- Adult Control (No Intervention): No intervention.

INTERVENTIONS:
Other: Pediatric Moisturizer — Apply moisturizer for four weeks daily to only one arm. Do not apply moisturizer to the other arm.
  Other Names: Cetaphil Cream; Aveeno Eczema Therapy Moisturizing Cream; CeraVe Moisturizing Cream; Aveeno Skin Relief Moisture Repair Cream
  Arms: Pediatric Moisturizer Intervention
Other: Adult Moisturizer — Apply moisturizer for four weeks daily to only one arm. Do not apply moisturizer to the other arm.
  Other Names: Cetaphil Cream; Aveeno Eczema Therapy Moisturizing Cream; CeraVe Moisturizing Cream; Vaseline 100% Petroleum Jelly
  Arms: Adult Moisturizer Intervention

SUMMARY:
The goal of this study is to better understand what effect emollients (moisturizers) have on the skin in young children and adults.

Subjects will be recruited from PI and Sub-I clinics and Oregon Health & Science University (OHSU) research opportunities website.

1. Adult and Adolescent Study:

   Moisturizer Intervention - There will be 2-3 visits for this study: a screening visit, a baseline visit, and a final visit. Adults with a history of eczema will be asked to apply one of four possible moisturizers to one arm and nothing to the other arm for four weeks. The moisturizers, which will be assigned to the subjects, include either Cetaphil Cream, Aveeno Eczema Therapy Moisturizing Cream, CeraVe Moisturizing Cream, or Vaseline 100% Petroleum Jelly. Subjects can use other skin treatments as needed for their skin condition, but may not treat the arms during the study. Non-invasive tests of the skin will be made at Visit 1 and after four weeks (Visit 2). The skin measurements that will be performed are:
   * Transepidermal loss (TEWL)- measures how much water is lost across the skin barrier
   * Skin Cohesion and TEWL - TEWL after 5, 10, 15, and 20 tape strips will measure skin barrier function after tape-stripping
   * Skin electrical capacitance - measures the moisture in the top layer of skin
   * Skin pH - measures the acidity of the skin
   * Stratum corneum cohesion assay - tape-stripping to measure the protein removed from the top layer of skin
   * Lipidomic analysis - measures the lipids, or oils, in the top layer of skin Control - There will be 1-2 visits for this group: a screening visit and baseline visit, which can be combined. Non-invasive tests of the skin will be taken and include the skin measurements that will be performed are the same as the Moisturizer Intervention group.
2. Pediatric Study: There will be 2-3 visits for this study: a screening visit, a baseline visit, and a final visit. Infants and toddlers between 3 months and 3 years of age without a history of skin barrier diseases will be assigned to a moisturizer, which include either Cetaphil Cream, Aveeno Eczema Therapy Moisturizing Cream, CeraVe Moisturizing Cream, or Aveeno Skin Relief Moisture Repair Cream. Non-invasive tests of the skin will be made at Visit 1 and after four weeks (Visit 2).

   * TEWL- measures how much water is lost across the skin barrier
   * Skin electrical capacitance - measures the moisture in the top layer of skin
   * Skin pH - measures the acidity of the skin

ELIGIBILITY:
1. Pediatric study

   * Inclusion Criteria

     * Enrollment in the BEEP emollient intervention study (IRB #6083)
     * Overall good health
   * Exclusion Criteria

     * Have a history of or are being evaluated for a skin barrier disease
     * Have an active skin infection
     * Are receiving phototherapy
     * Any immunodeficiency disorder or severe genetic skin disorder
     * Any other serious condition that would make the use of emollients inadvisable
     * Any other major medical problems that the investigator deems may increase the risk of adverse events with the intervention
2. Adult Study

   * Inclusion Criteria

     * Have a history of atopic dermatitis
     * 12 years or older
     * 4 x 4 cm of non-lesional skin on both inner forearms
     * No other conditions that would make the use of the four emollients harmful to the subject, such as known allergy to an emollient or a component o the emollient
   * Exclusion Criteria

     * Use of topical steroids on the inner forearms or oral immunosuppressive medications for 4 weeks prior to participation in the study.
     * Receiving phototherapy or systemic immunosuppressive therapy three months prior to participation in the study.

Ages: 3 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with improved skin barrier function as a result of emollient use | 3-4 weeks
  Change in TEWL measurements of intervention arms compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Simpson, MD, MCR, Principal Investigator — Oregon Health & Science University, Department of Dermatology
Locations (1):
- Oregon Health & Science University Center for Health & Healing, Portland, Oregon, United States